CLINICAL TRIAL: NCT07139067
Title: Phase I Clinical Study of YK1101 Injection for the Treatment of Advanced Solid Tumors
Acronym: YK1101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Yingkai Saiwei（Beijing）Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YK1101
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor Cancer
Keywords: Biological: TCR-T therapy; Phase I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YK1101 cells (Experimental): Biological: YK1101 cells Drug: Fludarabine + Cyclophosphamide
  Interventions: Biological: YK1101 cells

INTERVENTIONS:
Biological: YK1101 cells — Drug: Fludarabine + Cyclophosphamide

SUMMARY:
A single-arm, open-label, dose exploratory study to evaluate the safety, efficacy, and pharmacokinetics of autologous humanized anti-MAGE-A4 T cell receptor-engineered T cell (TCR-T) in advanced solid tumors.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, dose escalation/dose regimen finding study to assess the safety and pharmacokinetics of T-cell receptor-engineered T cell (TCR-T) targeting melanoma-associated antigen-4 (MAGE-A4) and to obtain the preliminary efficacy results in subjects who have been diagnosed with advanced solid tumors with positive MAGE-A4 expression.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily willing to participate in the study and sign the written informed consent form
2. Age ≥18 years and ≤75 years,male or female .
3. Human leukocyte antigen (HLA)-A*11:01 matched
4. Fresh or formalin-fixed paraffin-embedded (FFPE) samples, immunohistochemistry(IHC)-stained MAGE-A4 positive（+2，≥30%）
5. Histologically-confirmed recurrent/metastatic advanced solid tumors，have failed or relapsed with the standard regimen, or have not tolerated the standard treatment regimen.Including but not limited to synovial sarcoma, myxoid liposarcoma, urothelial carcinoma, esophagogastric junction carcinoma, ovarian carcinoma, esophageal squamous carcinoma, head and neck tumor, non-small cell lung squamous carcinoma, triple negative breast cancer, etc.
6. Patients must have at least one measurable lesion defined by RECIST 1.1.
7. No systemic anti-tumor therapy received within 2 weeks prior to peripheral blood mononuclear cell (PBMC) collection.
8. European Cooperative Oncology Group (ECOG) ≤1 and expected survival time ≥3 months at screening, 24 hours prior to apheresis (APH), lymphodepletion (LD), and infusion
9. Blood oxygen saturation (finger oxygen detection)≥ 95% in a calm and non oxygenated state.
10. Patients must meet the following criteria at screening and before preconditioning (baseline). If any laboratory test result is abnormal referring to the following criteria, it is acceptable to test one more time within 1week. If the test result is still abnormal, the patient is screen failed:

1）Hematology (no intensive blood transfusion (≥2 times within 1week), platelet transfusion or cell growth factor (except for recombinant erythropoietin) performed within 7days before the test): neutrophils (NE) ≥1.5×109 per liter, lymphocytes (LY) ≥0.5×109per liter (except for before preconditioning), platelets (PLT) ≥75×109per liter and hemoglobin (Hb) ≥8.0 g/dL.

2）Blood chemistry: creatinine clearance ≥40 mL/min, alanine aminotransferase (ALT) ≤2.5×ULN, aspartate aminotransferase (AST) ≤2.5×ULN, total bilirubin (TB) ≤1.5×ULN（Gilbert syndrome or liver metastasis subjects ≤ 3 × ULN）, serum lipase and amylase <1.5 ULN, alkaline phosphatase (ALP) ≤2.5 ULN; for patients with bone or hepatic metastasis, AST, ALT and ALP <5ULN.

3）Prothrombin time ≤ULN+4 seconds. 11. Women of childbearing potential must have negative serum pregnancy test result at screening and before preconditioning and agree to use an effective and reliable contraceptive method for at least 1 year after the last study treatment. Te acceptable methods include bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusion; any approved oral, injection or implantation of hormone; or barrier contraceptive method: condoms containing spermicidal .

Exclusion Criteria:

1. Pregnant or lactating women.
2. HIV, treponema pallidum or HCV serology is positive.
3. Patients with any uncontrolled active infection, including, but not limited to, active tuberculosis or HBV infection (HBsAg positive or HBV DNA positive).
4. Patients with symptomatic central nervous metastases.
5. Patients with AEs induced by previous treatment that have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤1, except for alopecia and other tolerable events judged by the investigator or permitted laboratory abnormalities according to the protocol.
6. Patient allergic or intolerant to preconditioning drugs, including, but not limited to, fudarabine and cyclophosphamide ; allergic to the components of YK1101; penicillin allergy history confrmed by positive skin test; or any severe allergy history-for example, anaphylactic shock.
7. Patients who have undergone coronary artery reconstruction in the past.
8. The patient's tumor lesion invades large blood vessels and has a significant risk of bleeding.
9. Thrombosis and embolism occurred 6 months before cell transfusion.
10. Patients who have undergone major surgery or severe trauma within 4weeks before apheresis .
11. Patients who have a history of organ transplantation or are waiting for organ transplantation.
12. Patients with other serious diseases that may restrict them from participating in this study, such as poorly controlled diabetes (glycosylated hemoglobin HbA1c >8% undertreatment), poorly controlled hypertension judged by the investigator (blood pressure >160mmHg/100mmHg), severe cardiac insufficiency (left ventricular ejection fraction <50%), myocardial infarction or unstable arrhythmia or unstable angina pectoris, pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease or clinically significant lung function test abnormalities in the past 6months.
13. Patients who are expected to continue using immunosuppressive therapy during the trial (excluding physiological replacement therapy with glucocorticoids, such as prednisone<10mg/d or equivalent doses)
14. Patients who require long-term use of aspirin or anticoagulant drugs.
15. Patients who have participated in other intervention clinical trials within 2 weeks.
16. Patients with adverse drug addiction or a history of drug abuse.
17. Patients who are unable or unwilling to comply with the clinical protocol, by the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
  Dose-limiting toxicity
Treatment related AEs | 28 days
  Treatment related AEs

SECONDARY OUTCOMES:
Antitumor efficacy-Objective response rate (ORR) | 2 years
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%).
Antitumor efficacy-Progression-free survival (PFS) | 2 years
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first.
Antitumor efficacy-Overall survival (OS) | 2 years
  The period from the first infusion to any cause of death
Antitumor efficacy-Duration of response (DOR) | 2 years
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of GI Oncology, Peking University Cancer Hospital Recruiting Beijing, Beijing, China, 100142, Beijing
  - Peking University Cancer Hospital & Institute, Beijing

IPD SHARING:
Plan to Share IPD: No